CLINICAL TRIAL: NCT04135638
Title: Comparing Retinal Sensitivity and Fixation Stability of Inverted ILM-flap Techniques Variants for Macular Hole Surgery
Brief Title: Inverted ILM-flap Techniques Variants for Macular Hole Surgery: Outcomes Comparison
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Molise (Other)
Collaborators: Ospedale Policlinico San Martino (Other); Fondazione G.B. Bietti, IRCCS (Other); Università degli Studi 'G. d'Annunzio' Chieti e Pescara (Other)
Responsible Party: Principal Investigator, Ciro Costagliola, Full Professor in Ophthalmology, University of Molise
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 14738
Record Dates: First submitted 2019-10-04; First posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Macular Holes
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cover Group (CG) (Other): All patients will undergo a 25G standard 3-port PPV with posterior vitreous detachment induction (if not already present), ILM staining with 0,25 g/l of brilliant blue-G and creation of a 360°ILM flap around the MH rim.
  Phakic patients will undergo combined phacoemulsification with IOL implant in-the-bag.
  In the Cover Group the ILM flap will be folded as a single layer to bridge tissue dehiscence during air-fluid exchange. All eyes will recive a mixture of 20% sulfur hexafluoride tamponade and will be instructed to position face down for 4 hours a day during the first 3 days post-operative
  Interventions: Procedure: Cover Group
- Fill Group (FG) (Other): All patients will undergo a 25G standard 3-port PPV with posterior vitreous detachment induction (if not already present), ILM staining with 0,25 g/l of brilliant blue-G and creation of a 360°ILM flap around the MH rim.
  Phakic patients will undergo combined phacoemulsification with IOL implant in-the-bag.
  In the Fill Group, multiple layers of ILM will be deliberately folded within the loss of tissue before air-fluid exchange. All eyes will receive a mixture of 20% sulfur hexafluoride tamponade and will be instructed to position face down for 4 hours a day during the first 3 days post-operative
  Interventions: Procedure: Fill Group

INTERVENTIONS:
Procedure: Cover Group — "Cover" when the ILM flap is everted over the MH gap in a single layer
  Arms: Cover Group (CG)
Procedure: Fill Group — "Fill" when the ILM is folded into multiple layers within the MH
  Arms: Fill Group (FG)

SUMMARY:
To report closure rate, Best Corrected Visual Acuity (BCVA), Retinal Sensitivity (RS) and Fixation Stability (FS) of idiopathic Macular Holes (MH) randomized to Cover Group (CG) or Fill Group (FG) of the Inverted Internal Limiting Membrane (ILM) flap surgical procedure.

DETAILED DESCRIPTION:
Patients will be randomized (1:1) to receive a vitrectomy with either Cover or Fill ILM flap technique. "Cover" when the ILM flap is everted over the MH gap in a single layer, "Fill" when the ILM is folded into multiple layers within the MH. All patients will undergo BCVA, RS and FS assessment at baseline, 1-month and 3-months after surgery.

Purpose of the study is to report retinal differential sensitivity and fixation stability as well as anatomic and visual outcomes of patients operated on for idiopathic MH and randomly assigned to Fill or Cover Groups.

ELIGIBILITY:
Inclusion Criteria:

* patients with idiopatic macular holes

Exclusion Criteria:

* Patients with MH duration greater than 6 months
* myopia exceeding 6 diopters
* history of trauma
* previous ocular surgery except uncomplicated cataract extraction with in-the-bag IOL implantation
* any ocular illness including glaucoma, uveitis, optic nerve pathology

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-04-10 (Estimated)

PRIMARY OUTCOMES:
Visual outcome linked to "Cover" and "Fill" procedures | five months
  To report :
  - Best Corrected Visual Acuity (BCVA expressed in logMAR)
  of idiopathic Macular Holes (MH) randomized to Cover Group (CG) or Fill Group (FG) of the Inverted Internal Limiting Membrane (ILM) flap surgical procedure.
Anatomical outcome linked to "Cover" and "Fill" procedures | five months
  To report:
  - closure rate (μm)
  of idiopathic Macular Holes (MH) randomized to Cover Group (CG) or Fill Group (FG) of the Inverted Internal Limiting Membrane (ILM) flap surgical procedure

SECONDARY OUTCOMES:
Macular sensitivity linked to "Cover" and "Fill" procedures | five months
  To report:
  * Retinal Sensitivity (RS expressed in dB)
  * Fixation Stability (FS expressed as: 0 = stable, 1 = relatively (stable,2 = unstable)
  of idiopathic Macular Holes (MH) randomized to Cover Group (CG) or Fill Group (FG) of the Inverted Internal Limiting Membrane (ILM) flap surgical procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Ciro Costagliola, Principal Investigator — University of Molise
Locations (1):
- University of Molise, Campobasso, Italy

REFERENCES:
- [Background] Kelly NE, Wendel RT. Vitreous surgery for idiopathic macular holes. Results of a pilot study. Arch Ophthalmol. 1991 May;109(5):654-9. doi: 10.1001/archopht.1991.01080050068031. PMID 2025167
- [Background] Michalewska Z, Michalewski J, Adelman RA, Nawrocki J. Inverted internal limiting membrane flap technique for large macular holes. Ophthalmology. 2010 Oct;117(10):2018-25. doi: 10.1016/j.ophtha.2010.02.011. Epub 2010 Jun 11. PMID 20541263
- [Background] Rossi T, Gelso A, Costagliola C, Trillo C, Costa A, Gesualdo C, Ripandelli G. Macular hole closure patterns associated with different internal limiting membrane flap techniques. Graefes Arch Clin Exp Ophthalmol. 2017 Jun;255(6):1073-1078. doi: 10.1007/s00417-017-3598-9. Epub 2017 Feb 4. PMID 28161828
- [Background] Molina-Martin A, Perez-Cambrodi RJ, Pinero DP. Current Clinical Application of Microperimetry: A Review. Semin Ophthalmol. 2018;33(5):620-628. doi: 10.1080/08820538.2017.1375125. Epub 2017 Oct 9. PMID 28991503
- [Background] Chen WC, Wang Y, Li XX. Morphologic and functional evaluation before and after successful macular hole surgery using spectral-domain optical coherence tomography combined with microperimetry. Retina. 2012 Oct;32(9):1733-42. doi: 10.1097/IAE.0b013e318242b81a. PMID 22466479
- [Background] Bonnabel A, Bron AM, Isaico R, Dugas B, Nicot F, Creuzot-Garcher C. Long-term anatomical and functional outcomes of idiopathic macular hole surgery. The yield of spectral-domain OCT combined with microperimetry. Graefes Arch Clin Exp Ophthalmol. 2013 Nov;251(11):2505-11. doi: 10.1007/s00417-013-2339-y. Epub 2013 Apr 26. PMID 23620091
- [Background] Chen SN. Large semicircular inverted internal limiting membrane flap in the treatment of macular hole in high myopia. Graefes Arch Clin Exp Ophthalmol. 2017 Dec;255(12):2337-2345. doi: 10.1007/s00417-017-3808-5. Epub 2017 Oct 10. PMID 28993905
- [Background] Aurora A, Seth A, Sanduja N. Cabbage Leaf Inverted Flap ILM Peeling for Macular Hole: A Novel Technique. Ophthalmic Surg Lasers Imaging Retina. 2017 Oct 1;48(10):830-832. doi: 10.3928/23258160-20170928-08. PMID 29020427
- [Background] Rizzo S, Tartaro R, Barca F, Caporossi T, Bacherini D, Giansanti F. INTERNAL LIMITING MEMBRANE PEELING VERSUS INVERTED FLAP TECHNIQUE FOR TREATMENT OF FULL-THICKNESS MACULAR HOLES: A COMPARATIVE STUDY IN A LARGE SERIES OF PATIENTS. Retina. 2018 Sep;38 Suppl 1:S73-S78. doi: 10.1097/IAE.0000000000001985. PMID 29232338
- [Background] Wang Z, Qi Y, Liang X, Yu Y, Chen J, Wang J, Liu X, Liu W. MP-3 measurement of retinal sensitivity in macular hole area and its predictive value on visual prognosis. Int Ophthalmol. 2019 Sep;39(9):1987-1994. doi: 10.1007/s10792-018-1032-x. Epub 2018 Oct 3. PMID 30284091
- [Background] Sun Z, Gan D, Jiang C, Wang M, Sprecher A, Jiang AC, Xu G. Effect of preoperative retinal sensitivity and fixation on long-term prognosis for idiopathic macular holes. Graefes Arch Clin Exp Ophthalmol. 2012 Nov;250(11):1587-96. doi: 10.1007/s00417-012-1997-5. Epub 2012 Mar 24. PMID 22441811
- [Background] Tarita-Nistor L, Gonzalez EG, Mandelcorn MS, Lillakas L, Steinbach MJ. Fixation stability, fixation location, and visual acuity after successful macular hole surgery. Invest Ophthalmol Vis Sci. 2009 Jan;50(1):84-9. doi: 10.1167/iovs.08-2342. Epub 2008 Aug 29. PMID 18757517
- [Derived] Cacciamani A, Gelso A, Di Nicola M, Scarinci F, Ripandelli G, Costagliola C, Rossi T. Inverted ILM-flap techniques variants for macular hole surgery: randomized clinical trial to compare retinal sensitivity and fixation stability. Sci Rep. 2020 Sep 28;10(1):15832. doi: 10.1038/s41598-020-72774-1. PMID 32985592